CLINICAL TRIAL: NCT06873971
Title: Effects of Erbium:YAG Laser Combined With Vaginal Estriol Therapy in Postmenopausal Women With Genitourinary Syndrome of Menopause: A Protocol for a Randomised, Double-blind Controlled Trial
Brief Title: Er:YAG Laser Combined With Vaginal Estriol for Genitourinary Syndrome of Menopause
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Stella Regina Zamuner, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERBIUM-YAG-LASER
Record Dates: First submitted 2025-02-21; First posted 2025-03-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: Genitourinary syndrome of menopause; postmenopausal women; Erbium: YAG laser; vaginal microbiome; vaginal estriol
MeSH Terms: interventions — Estriol; Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Vaginal estriol plus Sham Er:YAG laser (minimal fluence)) (Sham Comparator): All participants will receive vaginal estriol therapy combined with Er:YAG laser intervention with minimal fluence (0.5 J/cm²), below the threshold for biological tissue effect, applied to maintain participant blinding through auditory and procedural cue. Participants will undergo three laser applications at four-week intervals. The intimate laser session consists of two stages using a PS03 fractional tip: the internal stage (vaginal canal) with energy settings of 0.5 J/cm² at 2 Hz, and the external stage (vulvar and vestibule region) with energy settings of 0.5J/cm² at 2 Hz.
  Interventions: Drug: Topical estrogen therapy based on estriol (E3); Radiation: Sham Er:YAG laser (minimal fluence)
- GROUP 2 ( Vaginal estriol plus active Er:YAG laser) (Active Comparator): All participants will receive vaginal estriol therapy combined with an active Er:YAG (λ = 2940 nm) . Participants will undergo three laser applications at four-week intervals. The intimate laser session consists of two stages using a PS03 fractional tip: the internal stage (vaginal canal) with energy settings of 9 J/cm² at 2 Hz, and the external stage (vulvar and vestibule region with energy settings of 6 J/cm² at 2 Hz.The laser device to be used is the Smooth XS Dynamics Dualis (FOTONA, Ljubljana, Slovenia) with a wavelength of 2940 nm.
  Interventions: Drug: Topical estrogen therapy based on estriol (E3); Radiation: Active Er:YAG Laser

INTERVENTIONS:
Drug: Topical estrogen therapy based on estriol (E3) — All participants will use low-dose Vaginal estriol cream (1 mg/g) administered intravaginally using disposable, individualized vaginal applicators pre-set at the recommended dosage of 0.5g/ per application (equivalent to 0.5 mg of estriol per dose).
  Induction phase: 0.5 g once daily at bedtime for 14 consecutive days. Maintenance phase: 0.5 g twice weekly for 16 weeks, on Mondays and Thursdays. The treatment will be provided in fractions for each 30 day period and will always be delivered after each laser session, along with a leaflet containing usage, storage, and application instructions for the vaginal cream. The patients will be monitored through a messaging app, reinforcing the instructions and the days of application correctly.
  Other Names: Estriol ( E3); Vaginal estriol ( E3)
Radiation: Active Er:YAG Laser — All participants in the group will undergo 3 applications of active Er:YAG laser with an interval of 4-5 weeks between them. The intimate laser session consists of two stages using a PS03 fractional tip: the internal stage (vaginal canal) with energy settings of 9 J/cm² at 2 Hz, and the external stage (vulvar and vestibule region) with energy settings of 6 J/cm² at 2 Hz.The laser device to be used is the Smooth XS Dynamics Dualis (FOTONA, Ljubljana, Slovenia) with a wavelength of 2940 nm.
  Other Names: Laser On; Laser in Active Intervention Mode
  Arms: GROUP 2 ( Vaginal estriol plus active Er:YAG laser)
Radiation: Sham Er:YAG laser (minimal fluence) — All participants in the group will undergo 3 sham applications of Sham Er:YAG laser intervention delivered at minimal fluence (0.5 J), below the threshold for biological tissue effect, applied to preserve participant blinding through auditory and procedural cues , with an interval of 4-5 weeks between them. The intimate laser session consists of two stages using a PS03 fractional tip: the internal stage (vaginal canal) with energy settings of 0.5 J/cm² at 2 Hz, and the external stage (vestibule and introitus region) with energy settings of 0.5 J/cm² at 2 Hz.The laser device to be used is the Smooth XS Dynamics Dualis (FOTONA, Ljubljana, Slovenia) with a wavelength of 2940 nm.
  Other Names: Laser in Minimal Fluence
  Arms: GROUP 1 (Vaginal estriol plus Sham Er:YAG laser (minimal fluence))

SUMMARY:
Chronic hypoestrogenism in postmenopausal women significantly impacts the urogenital epithelium, leading to Genitourinary Syndrome of Menopause (GSM) and increasing susceptibility to gynecological infections due to vaginal pH elevation. Therapies using the Erbium:YAG (Er:YAG) 2940nm laser and low dose topical estrogen have demonstrated efficacy in improving vaginal trophism and restoring microbiota balance.

This randomised, double-blind clinical study aims to assess the effects of combining Er: YAG laser therapy with vaginal estriol compared with estriol therapy alone in postmenopausal women with GSM. Sixty patients will be recruited and randomly assigned to two groups. All participants will receive low-dose topical estrogen therapy (estriol cream ) for 14 days, followed by twice-weekly applications until completing three laser sessions at four-week intervals. Group 1 (Sham) will receive the laser with minimal fluence (0.5J/cm²) applied to maintain blinding (auditory cues) below the threshold for biological tissue, while Group 2 , will undergo active laser treatment.

Inclusion criteria include age 45-70 years, vaginal pH ≥5, absence of hormone therapy or energy-based intimate treatments for 180 days, and moderate vaginal atrophy symptoms (SCORE >4). Exclusion criteria include abnormal cervicalvaginal cytology in the last six months, corticosteroid therapy within 90 days, and BMI ≥35kg/m².

Assessments will occur at Baseline, 30 days after each laser session and 4 months after the third laser application. The primary outcome is the Vaginal Health Index (VHI), while secondary outcomes include GSM symptom evaluation via the Visual Analog Scale, vaginal microbiota analysis through 16S gene sequencing, and quality-of-life and sexual health questionnaires. Statistical analysis of the groups will be performed using SPSS version 22.0. For analytical statistics, repeated measures ANOVA will be used for continuous data, and non-parametric tests for repeated measures, such as the Friedman test, when appropriate. A p-value <0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Chronic, progressive hypoestrogenism, without adequate treatment during the postmenopausal period, significantly affects the epithelium of the urogenital system, causing Genitourinary Syndrome of Menopause (GSM). This disorder impacts the quality of life of thousands of women, favoring the emergence of other pathologies, including increasing the risk of gynecological infections from opportunistic microorganisms due to the elevation of vaginal pH, destabilizing the natural immunological barrier. Therapies using the Erbium:YAG (Er:YAG) 2940nm laser and low-dose topical estrogen therapy have demonstrated safety and efficacy in improving vaginal trophism, being crucial for the reestablishment of appropriate flora.

This study aims to assess the effects of combining Er: YAG laser therapy with vaginal estriol compared with estriol therapy alone in postmenopausal women with GSM. This is a randomised, double-blind clinical study. Sixty patients will be recruited and randomly divided into two groups. All participants will receive low-dose topical estrogen therapy (vaginal estriol cream (1 mg/g) administered intravaginally using disposable applicators pre-set to deliver 0.5 g per application (equivalent to 0.5 mg of estriol per dose) for 14 consecutive days and then twice weekly until completing three sessions of laser treatment, with a 4-week interval between sessions. In Group 1 (Sham), the laser will be applied with minimal fluence (0.5 J/cm²) to maintain blinding (auditory cues) below the threshold for biological tissue, while in Group 2, will be applied an active Er:YAG laser intervention. The intimate laser session consists of two stages: the internal stage ( vaginal canal) with energy settings of 9J/cm² at 2Hz and the external stage (vulvar and vestibule region) with energy settings of 6J/cm² at 2Hz.

Inclusion criteria include age between 45 and 70 years, vaginal pH level ≥5, absence of hormone therapy and intimate treatments using energy for 180 days, and presence of moderate symptoms of vaginal atrophy (SCORE >4). Exclusion criteria include altered cervical-vaginal cytology in the last six months, corticosteroid therapy within the last 90 days, and BMI ≥35kg/m².

Comparisons between the two groups will be conducted at Baseline, 30 days after each laser session and 4 months after the third laser application. The primary outcome will be the Vaginal Health Index (VHI). Secondary outcomes will include the Visual Analog Scale for four symptoms of GSM (burning, irritation, dyspareunia, and persistent leukorrhea), vaginal microbiological sampling for DNA sequencing analysis using the 16S gene amplification technique, specifically at the V3/V4 region (before the first laser therapy session and 4 weeks after the third application), quality of life, and sexual health questionnaires.

Data will be collected using coded identifiers and stored on a secure, password-protected institutional server with restricted access. Regular data backups will be performed. Only authorised members of the research team will have access to identifiable data. De-identified data may be shared upon reasonable request, subject to ethical approval and data-sharing agreements.

Statistical analysis of the groups will be performed using SPSS version 22.0. For analytical statistics, repeated measures ANOVA will be used for continuous data, and non-parametric tests for repeated measures, such as the Friedman test, when appropriate. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria

* Postmenopausal women (45-70 years of age).
* At least one of moderate symptom of GSM (vaginal dryness, burning sensation, dyspareunia, and persistent leukorrhea), defined by ≥ 4 on Visual Analog Scale (VAS) ranging from 0 to 10.
* Vaginal pH ≥5.0 at baseline assessment.
* Not having undergone hormone replacement therapy (vaginal or systemic) in the previous six months.
* No use of vaginal moisturizers in the previous 30 days.
* Demonstrated capacity and willingness to provide written informed consent and adhere to study protocols.

Exclusion criteria

* Vaginal or vulvar energy-based interventions (e.g., laser, radiofrequency) in the previous six months.
* Abnormal cervical cytology, specifically ASCUS, LSIL, or HSIL, documented in the previous six months.
* Systemic corticosteroid therapy administered in the previous 90 days.
* Body mass index (BMI) ≥35 kg/m².
* Presence of abnormal uterine bleeding in the previous 30 days.
* History of vaginal surgery in the previous 180 days or grade II or higher uterine prolapse (POP-q).
* History of malignant neoplasms or exposure to vaginal radiotherapy.
* Diagnosis of severe liver or kidney disease, autoimmune disease, or severe psychiatric disorder.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of the Vaginal Health Index (VHI) | Baseline, 30 days after each laser session and 4 months after the third laser application.
  Clinically assesses the degree of genital atrophy through physical examination, which analyzes "urogenital health." This is useful for the longitudinal follow-up of patients, where changes occurring in the genitourinary tract are noted, including the analysis of the need for therapeutic intervention. The parameters analyzed are: total elasticity, type and consistency of fluid secretion, Vaginal pH, epithelial mucosa, and moisture, which, according to their characteristics, receive scores from 1 to 5. The lower the score, the greater the degree of urogenital atrophy.
  Vaginal pH will be assessed as an integral component of the Vaginal Health Index and will not be analysed as a separate outcome measure.

SECONDARY OUTCOMES:
Vaginal Microbiome | Before first laser session and four weeks after the third laser application.
  The analytical methodology involves sequencing the 16S rRNA gene (V3/V4) after DNA extraction using the "ZymoBIOMICS DNA Miniprep" kit, following the manufacturer's guidelines provided by "Biomehub Research and Development S.A." For bacterial identification, library preparation will be performed through amplification of the V3/V4 regions (341F and 806R) using a two-step PCR. The first PCR employs universal oligonucleotides for the V3/V4 region, while the second incorporates sequencing indexes. Sample collection will be conducted individually by the responsible researcher before the first laser session and four weeks after the third application. Statistical evaluations will include descriptive analysis, alpha diversity, beta diversity, and differential abundance between groups. Samples will be stored for three months and subsequently discarded by the contracted laboratory, adhering to the manufacturer's recommendations.
Visual Analog Scale (VAS) | baseline, 30 days after each laser session and four months after the third laser application
  Four types of symptoms of GSM (dryness, burning, dyspareunia, and chronic leukorrhea) will be evaluated separately by the patient according to the VAS criteria, ranging from 0 (absence of symptoms) to 10 (very severe symptoms). Moderate symptoms will be considered with values equal to or greater than 4.
Quality of Life Evaluation Questionnaires: Menopause Rating Scale (MRS) | Baseline, 30 days after each laser session and 4 months after the third laser application.
  Used to assess quality of life and symptoms related to climacteric. It consists of 11 questions distributed to analyze three parameters: somato-vegetative symptoms, psychological symptoms, and urogenital symptoms, which are classified into five degrees: none, mild, moderate, severe, and extremely severe. The higher the score, the greater the severity of the symptoms and, consequently, the worse the quality of life for the woman during the climacteric.
Female Sexual Function Index (FSFI) | Baseline, 30 days after each laser session and 4 months after the third laser application.
  A tool used to evaluate female sexual response, based on the analysis of six domains: sexual desire, sexual arousal, vaginal lubrication, orgasm, sexual satisfaction, and pain. This assists in understanding how various factors, including health, relationships, and psychosocial factors, influence sexual satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil